CLINICAL TRIAL: NCT03264001
Title: Effects of Progressive Negative Energy Balance Induced by Diet or Exercise on Glucose Tolerance, Insulin Sensitivity, and Beta-cell Function
Brief Title: Effects of Progressive Negative Energy Balance on Glucose Tolerance, Insulin Sensitivity, and Beta-cell Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Faidon Magkos, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEB
Record Dates: First submitted 2017-08-18; First posted 2017-08-28 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Insulin Sensitivity; Glucose Intolerance; Insulin Resistance; Energy Supply; Deficiency
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet-induced negative energy balance (Experimental): For the diet-induced negative energy balance arm, the three trials will include one control trial (isocaloric diet; zero energy balance) and two trials of progressively increasing negative energy balance induced by calorie restriction (20% and 40% reduction of daily energy needs for weight maintenance). With respect to physical activity, all diet trials will be performed under resting conditions.
  Interventions: Behavioral: Negative energy balance
- Exercise-induced negative energy balance (Experimental): For the exercise-induced negative energy balance arm, the three trials will include one control trial (rest; zero energy balance) and two trials of progressively increasing negative energy balance induced by aerobic exercise (20% and 40% reduction of daily energy needs for weight maintenance); with respect to caloric intake, all exercise trials will be performed under isocaloric conditions.
  Interventions: Behavioral: Negative energy balance

INTERVENTIONS:
Behavioral: Negative energy balance — 20% and 40% reduction of daily energy needs for weight maintenance

SUMMARY:
Type 2 diabetes results from a combination of peripheral insulin resistance and beta-cell dysfunction, and manifests as fasting and postprandial hyperglycemia. In Singapore, despite the relatively low prevalence of overweight and obesity, the prevalence of type 2 diabetes is disproportionately high and is expected to double in the near future. This indicates that insulin resistance and beta-cell dysfunction are widely prevalent even among individuals who are not overweight or obese. Still, weight loss induced by a variety of ways (calorie restriction, exercise, surgery, etc.) is considered the cornerstone of diabetes treatment. This underscores the importance of negative energy balance in improving metabolic function. In fact, negative energy balance induced by calorie restriction can improve metabolic function acutely, i.e. within 1-2 days and before any weight loss occurs. Likewise, negative energy balance induced by a single session of aerobic exercise improves metabolic function over the next few days. However, the magnitude of negative energy balance that needs to be achieved in order to improve metabolic function, as well as possible dose-response relationships, are not known. Furthermore, the comparative efficacy of calorie restriction vs. exercise in improving metabolic function has never been directly assessed.

Accordingly, a better understanding of the effects of acute negative energy balance induced by calorie restriction or aerobic exercise on insulin sensitivity and beta-cell function will have important implications for public health, by facilitating the design of effective lifestyle (diet and physical activity) interventions to prevent or treat type 2 diabetes.

To test these hypotheses, whole-body insulin sensitivity, the acute insulin response to glucose, and the disposition index (i.e. beta-cell function), will be determined the morning after a single day of progressively increasing negative energy balance (equivalent to 20% or 40% of total daily energy needs for weight maintenance) induced by calorie restriction or aerobic exercise.

Results from this project are expected to result in the better understanding of the effects of negative energy balance induced by diet and exercise on metabolic function. Therefore, this project may help in the design of effective lifestyle intervention programs for the prevention and treatment of type 2 diabetes.

DETAILED DESCRIPTION:
Metabolic dysfunction, obesity, and type 2 diabetes The incidence of overweight and obesity has been increasing during the past 2-3 decades in Singapore, and is expected to rise further in the future. By the year 2050, it is estimated that more than half of the population will be overweight or obese, defined as having a body mass index (BMI, calculated as the weight in kilograms divided by the square of height in meters) equal to or greater than 25 kg/m2. This is likely responsible, at least in part, for the concomitant increase in obesity-related co-morbid conditions, and particularly type 2 diabetes. The relationship between BMI and the risk for type 2 diabetes in populations from the Asia-Pacific region is linear within a wide range of BMI values (from ~21 kg/m2 to ~34 kg/m2), so that for every 2 kg/m2 increase in BMI (which corresponds to ~6 kg for a normal-weight person of average stature), the risk for developing type 2 diabetes rises by ~27 %. In Singapore, the prevalence of type 2 diabetes is expected to double from 7.3 % in 1990 to ~15 % in 2050, predominantly as a result of the fattening of the population. Remarkably, however, the prevalence of type 2 diabetes in Singapore is similar to that in the Unites States, even though the prevalence of overweight and obesity (BMI ≥25 kg/m2) is approximately half. This corroborates findings from many studies demonstrating that markers of metabolic dysfunction and particularly hyperglycemia, hyperinsulinemia, and insulin resistance, are highly prevalent among Singaporean adults, even among people who are not overweight or obese. This likely results in increased risk for developing type 2 diabetes. These observations underscore the importance of metabolic dysfunction independent of body weight per se.

Metabolic effects of weight loss The pathogenesis of type 2 diabetes involves peripheral insulin resistance (i.e. resistance of peripheral tissues and particularly skeletal muscle to the glucose uptake-promoting effect of insulin) and inadequate secretion of insulin from the pancreatic beta-cells upon glucose stimulation, leading to fasting and postprandial hyperglycemia. Weight loss, achieved as a result of chronic negative energy balance induced by a variety of ways (calorie restriction, exercise, pharmacotherapy, bariatric surgery), improves metabolic function and is considered the cornerstone of diabetes prevention and management. Part of the beneficial effect of weight loss could be due to the reduction in total body fat, intra-abdominal fat, and ectopic fat accumulation in metabolically active organs (e.g. muscle, pancreas, and liver), however acute perturbations in energy balance (whether positive or negative, for a period of 24-72 hours) can affect insulin action, beta-cell function, and glycemic control even before any changes in body weight or body fat distribution occur. For example, one day of overfeeding disrupts 24-hr glucose homeostasis, and two days of caloric restriction improves insulin action. Likewise, exercise can also lead to negative energy balance and is a very potent intervention that readily improves metabolic function and particularly insulin sensitivity, even after just a single session. Nevertheless, the degree of negative energy balance that needs to be achieved by calorie restriction or exercise in order to improve insulin action and beta-cell function is not known, and the dose-response relationship between negative energy balance and metabolic function remains elusive. Furthermore, the comparative efficacy of calorie restriction and exercise on improving the mechanisms regulating glucose homeostasis (i.e. insulin sensitivity and beta-cell function) has not been adequately studied. One study found that for the same amount weight loss (8-9 % of initial body weight) induced by a low-calorie diet or endurance exercise, exercise caused a greater reduction in fat mass, a smaller decrease in muscle mass, and led to a greater increase in insulin-mediated glucose disposal during a hyperinsulinemic-euglycemic clamp (by ~30 %), and a greater reduction in the total insulin response to an oral glucose tolerance test (by ~2.5-fold), compared with matched diet-induced weight loss; although these differences did not reach statistical significance. These observations raise the possibility that, for the same negative energy balance, exercise may be more effective than calorie restriction in improving metabolic function; however these findings are difficult to interpret in the face of the concomitant more favorable changes in body composition and fat distribution. No study has directly assessed the effects of the same acute negative energy balance induced by calorie restriction or aerobic exercise on metabolic function.

Accordingly, a better understanding of the effects of calorie restriction and exercise on insulin sensitivity, beta-cell function and daily glycemic control will have important implications for the design of effective lifestyle intervention targeted at preventing or managing type 2 diabetes. To this end, this study aims to test the following hypotheses:

Hypothesis 1: It is hypothesized that a single day of negative energy balance induced by calorie restriction improves intravenous glucose tolerance because of improved beta-cell function without changes in insulin sensitivity. The investigators further hypothesize that this effect requires 20% negative energy balance, and does not improve further with greater energy restriction (40%).

Hypothesis 2: It is hypothesized that a single day of negative energy balance induced by aerobic exercise improves intravenous glucose tolerance because of improved insulin sensitivity without changes in beta-cell function. The investigators further hypothesize this effect requires 20% negative energy balance, and improves further with greater energy restriction (40%).

Hypothesis 3: It is hypothesized that at any given level of negative energy balance (20% or 40%), calorie restriction has a greater effect than aerobic exercise on beta-cell function, whereas aerobic exercise has a greater effect than calorie restriction on insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Age between 21-65 years
* BMI from ≥18 to <30 kg/m2 (BMI is equal to body weight in kilograms divided by height in metres squared)

Exclusion Criteria:

* Persons with metabolic diseases that require use of medications (e.g. diabetes, heart disease, hypertension, etc.)
* Persons using tobacco products (smokes daily or occasionally)
* Persons who regularly consume alcohol (≥1 drink/day)
* Women on oral contraceptives or hormone replacement therapy
* Pregnant or breastfeeding women
* Persons who have had recent weight loss or gain (≥5% over the past 6 months)
* Persons with contraindication to calorie restriction (e.g. anemia) or exercise (e.g. asthma)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 4-6 weeks
  Insulin sensitivity index (i.e. Si) will be determined by using minimal modeling analysis of the IVGTT data.
Beta-cell function | 4-6 weeks
  Beta-cell function will be determined as the disposition index (i.e. product of acute insulin response [AIR] and Si) using minimal modeling analysis of the IVGTT data.

CONTACTS AND LOCATIONS:
Overall Officials: Faidon Magkos, PhD, Principal Investigator — Clinical Nutrition Research Centre
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phan TP, Alkema L, Tai ES, Tan KH, Yang Q, Lim WY, Teo YY, Cheng CY, Wang X, Wong TY, Chia KS, Cook AR. Forecasting the burden of type 2 diabetes in Singapore using a demographic epidemiological model of Singapore. BMJ Open Diabetes Res Care. 2014 Jun 11;2(1):e000012. doi: 10.1136/bmjdrc-2013-000012. eCollection 2014. PMID 25452860
- [Background] Asia Pacific Cohort Studies Collaboration; Ni Mhurchu C, Parag V, Nakamura M, Patel A, Rodgers A, Lam TH. Body mass index and risk of diabetes mellitus in the Asia-Pacific region. Asia Pac J Clin Nutr. 2006;15(2):127-33. PMID 16672195
- [Background] Yoon KH, Lee JH, Kim JW, Cho JH, Choi YH, Ko SH, Zimmet P, Son HY. Epidemic obesity and type 2 diabetes in Asia. Lancet. 2006 Nov 11;368(9548):1681-8. doi: 10.1016/S0140-6736(06)69703-1. PMID 17098087
- [Background] Deurenberg-Yap M, Yian TB, Kai CS, Deurenberg P, VAN Staveren WA. Manifestation of cardiovascular risk factors at low levels of body mass index and waist-to-hip ratio in Singaporean Chinese. Asia Pac J Clin Nutr. 1999 Sep;8(3):177-83. doi: 10.1046/j.1440-6047.1999.00091.x. PMID 24394159
- [Background] Deurenberg-Yap M, Chew SK, Lin VF, Tan BY, van Staveren WA, Deurenberg P. Relationships between indices of obesity and its co-morbidities in multi-ethnic Singapore. Int J Obes Relat Metab Disord. 2001 Oct;25(10):1554-62. doi: 10.1038/sj.ijo.0801739. PMID 11673781
- [Background] Luo D, Liu F, Li X, Yin D, Lin Z, Liu H, Hou X, Wang C, Jia W. Comparison of the effect of 'metabolically healthy but obese' and 'metabolically abnormal but not obese' phenotypes on development of diabetes and cardiovascular disease in Chinese. Endocrine. 2015 May;49(1):130-8. doi: 10.1007/s12020-014-0444-2. Epub 2014 Oct 14. PMID 25312689
- [Background] Bradley D, Magkos F, Klein S. Effects of bariatric surgery on glucose homeostasis and type 2 diabetes. Gastroenterology. 2012 Oct;143(4):897-912. doi: 10.1053/j.gastro.2012.07.114. Epub 2012 Aug 8. PMID 22885332
- [Background] Aucott L, Poobalan A, Smith WC, Avenell A, Jung R, Broom J, Grant AM. Weight loss in obese diabetic and non-diabetic individuals and long-term diabetes outcomes--a systematic review. Diabetes Obes Metab. 2004 Mar;6(2):85-94. doi: 10.1111/j.1462-8902.2004.00315.x. PMID 14746573
- [Background] Maggard-Gibbons M, Maglione M, Livhits M, Ewing B, Maher AR, Hu J, Li Z, Shekelle PG. Bariatric surgery for weight loss and glycemic control in nonmorbidly obese adults with diabetes: a systematic review. JAMA. 2013 Jun 5;309(21):2250-61. doi: 10.1001/jama.2013.4851. PMID 23736734
- [Background] Magkos F, Fraterrigo G, Yoshino J, Luecking C, Kirbach K, Kelly SC, de las Fuentes L, He S, Okunade AL, Patterson BW, Klein S. Effects of Moderate and Subsequent Progressive Weight Loss on Metabolic Function and Adipose Tissue Biology in Humans with Obesity. Cell Metab. 2016 Apr 12;23(4):591-601. doi: 10.1016/j.cmet.2016.02.005. Epub 2016 Feb 22. PMID 26916363
- [Background] Magkos F, Yannakoulia M, Chan JL, Mantzoros CS. Management of the metabolic syndrome and type 2 diabetes through lifestyle modification. Annu Rev Nutr. 2009;29:223-56. doi: 10.1146/annurev-nutr-080508-141200. PMID 19400751
- [Background] Gaborit B, Abdesselam I, Kober F, Jacquier A, Ronsin O, Emungania O, Lesavre N, Alessi MC, Martin JC, Bernard M, Dutour A. Ectopic fat storage in the pancreas using 1H-MRS: importance of diabetic status and modulation with bariatric surgery-induced weight loss. Int J Obes (Lond). 2015 Mar;39(3):480-7. doi: 10.1038/ijo.2014.126. Epub 2014 Jul 21. PMID 25042860
- [Background] Kirk E, Reeds DN, Finck BN, Mayurranjan SM, Patterson BW, Klein S. Dietary fat and carbohydrates differentially alter insulin sensitivity during caloric restriction. Gastroenterology. 2009 May;136(5):1552-60. doi: 10.1053/j.gastro.2009.01.048. Epub 2009 Jan 25. PMID 19208352
- [Background] Magkos F, Smith GI, Reeds DN, Okunade A, Patterson BW, Mittendorfer B. One day of overfeeding impairs nocturnal glucose but not fatty acid homeostasis in overweight men. Obesity (Silver Spring). 2014 Feb;22(2):435-40. doi: 10.1002/oby.20562. Epub 2013 Sep 10. PMID 23836730
- [Background] Thomas F, Smith GC, Lu J, Babor R, Booth M, Beban G, Chase JG, Murphy R. Differential Acute Impacts of Sleeve Gastrectomy, Roux-en-Y Gastric Bypass Surgery and Matched Caloric Restriction Diet on Insulin Secretion, Insulin Effectiveness and Non-Esterified Fatty Acid Levels Among Patients with Type 2 Diabetes. Obes Surg. 2016 Aug;26(8):1924-31. doi: 10.1007/s11695-015-2038-3. PMID 26729277
- [Background] Plourde CE, Grenier-Larouche T, Caron-Dorval D, Biron S, Marceau S, Lebel S, Biertho L, Tchernof A, Richard D, Carpentier AC. Biliopancreatic diversion with duodenal switch improves insulin sensitivity and secretion through caloric restriction. Obesity (Silver Spring). 2014 Aug;22(8):1838-46. doi: 10.1002/oby.20771. Epub 2014 Apr 24. PMID 24760439
- [Background] Magkos, F. and L.S. Sidossis, Exercise and insulin sensitivity. Where do we stand? You'd better run! European Endocrinology, 2008. 4(1): p. 22-25.
- [Background] Magkos F, Tsekouras Y, Kavouras SA, Mittendorfer B, Sidossis LS. Improved insulin sensitivity after a single bout of exercise is curvilinearly related to exercise energy expenditure. Clin Sci (Lond). 2008 Jan;114(1):59-64. doi: 10.1042/CS20070134. PMID 17635103
- [Background] Mikines KJ, Sonne B, Farrell PA, Tronier B, Galbo H. Effect of physical exercise on sensitivity and responsiveness to insulin in humans. Am J Physiol. 1988 Mar;254(3 Pt 1):E248-59. doi: 10.1152/ajpendo.1988.254.3.E248. PMID 3126668
- [Background] Ross R, Dagnone D, Jones PJ, Smith H, Paddags A, Hudson R, Janssen I. Reduction in obesity and related comorbid conditions after diet-induced weight loss or exercise-induced weight loss in men. A randomized, controlled trial. Ann Intern Med. 2000 Jul 18;133(2):92-103. doi: 10.7326/0003-4819-133-2-200007180-00008. PMID 10896648
- [Background] Weiss EP, Racette SB, Villareal DT, Fontana L, Steger-May K, Schechtman KB, Klein S, Holloszy JO; Washington University School of Medicine CALERIE Group. Improvements in glucose tolerance and insulin action induced by increasing energy expenditure or decreasing energy intake: a randomized controlled trial. Am J Clin Nutr. 2006 Nov;84(5):1033-42. doi: 10.1093/ajcn/84.5.1033. PMID 17093155
- [Background] Weir JB. New methods for calculating metabolic rate with special reference to protein metabolism. 1949. Nutrition. 1990 May-Jun;6(3):213-21. No abstract available. PMID 2136000
- [Background] Bergman RN, Ader M, Huecking K, Van Citters G. Accurate assessment of beta-cell function: the hyperbolic correction. Diabetes. 2002 Feb;51 Suppl 1:S212-20. doi: 10.2337/diabetes.51.2007.s212. PMID 11815482
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] Boston RC, Stefanovski D, Moate PJ, Sumner AE, Watanabe RM, Bergman RN. MINMOD Millennium: a computer program to calculate glucose effectiveness and insulin sensitivity from the frequently sampled intravenous glucose tolerance test. Diabetes Technol Ther. 2003;5(6):1003-15. doi: 10.1089/152091503322641060. PMID 14709204
- [Background] Ganda OP, Day JL, Soeldner JS, Connon JJ, Gleason RE. Reproducibility and comparative analysis of repeated intravenous and oral glucose tolerance tests. Diabetes. 1978 Jul;27(7):715-25. doi: 10.2337/diab.27.7.715. PMID 658617
- [Background] Prigeon RL, Kahn SE, Porte D Jr. Reliability of error estimates from the minimal model: implications for measurements in physiological studies. Am J Physiol. 1994 Feb;266(2 Pt 1):E279-86. doi: 10.1152/ajpendo.1994.266.2.E279. PMID 8141288
- [Derived] Tranaes K, Ding C, Chooi YC, Chan Z, Choo J, Leow MK, Magkos F. Dissociation Between Insulin Resistance and Abnormalities in Lipoprotein Particle Concentrations and Sizes in Normal-Weight Chinese Adults. Front Nutr. 2021 Feb 26;8:651199. doi: 10.3389/fnut.2021.651199. eCollection 2021. PMID 33718425
- [Derived] Ding C, Chooi YUC, Chan Z, Lo J, Choo J, Ding BTK, Leow MK, Magkos F. Dose-Dependent Effects of Exercise and Diet on Insulin Sensitivity and Secretion. Med Sci Sports Exerc. 2019 Oct;51(10):2109-2116. doi: 10.1249/MSS.0000000000002020. PMID 31033904